CLINICAL TRIAL: NCT05887505
Title: Effects of Vitamin D Status and Multiple Mega-dose Supplementation on Health Care Disparities in Perioperative Patients With Hepatocellular Carcinoma Receiving Hepatectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taoyuan General Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TYGH111086
Record Dates: First submitted 2023-05-02; First posted 2023-06-02 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-04

CONDITIONS: Hepatocellular Carcinoma; Liver Function; Postoperative Complications
Keywords: Vitamin D Supplementation; Hepatectomy; Perioperative
MeSH Terms: conditions — Carcinoma, Hepatocellular; Postoperative Complications | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D group (Experimental): Oral supplementation of 1,728,000 IU vitamin D3 in 3 days
  Interventions: Other: Vitamin D
- Placebo Group (Placebo Comparator): Oral supplementation of placebo in 3 days
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Vitamin D — Oral supplementation of 576,000IU/day vitamin D3 in 3 consecutive days
  Arms: Vitamin D group
Other: Placebo — Oral supplementation of placebo in 3 consecutive days.
  Arms: Placebo Group

SUMMARY:
High concentrations of parathyroid hormone (PTH) are common in patients with hepatocellular carcinoma (HCC). This study is aimed to investigate effects of vitamin D status and its multiple mega-dosage supplementation on PTH and clinical outcomes in HCC patients before and after hepatectomy. It's a single-center, prospective, parallel, double-blind, placebo-controlled study for 120 eligible subjects. The subjects will receive consecutively 3-day intervention treatments from 7th day before surgery. 30-day postoperative mortality, postoperative complications, and laboratory data will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 1. ≥ 20-year HCC subjects receiving laparoscopic hepatectomy
* 2.Sign the informed consent

Exclusion Criteria:

* 1. Using estrogen drugs, bisphosphonates, or drugs for bone disease.
* 2. Consume calcium tablets within 2 weeks before operation
* 3. Sarcoidosis, multiple myeloma
* 4. Pregnant women or plan to become pregnant within 3 months after surgery
* 5. Autoimmune hepatitis (AIH)
* 6. Early liver recurrence
* 7. Used to participate in other clinical trials

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-06-09 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Whether there is an association between 25(OH)D and PTH: positive or negative association , or no association | During the study period
Ratio of liver failure | 7 days pre- OP (day -7)
Ratio of liver failure | 1 day pre- OP (day -1)
Ratio of liver failure | 1 day post- OP (day 1)
Ratio of liver failure | 1 day before discharge

SECONDARY OUTCOMES:
25(OH)D status | Baseline (day -7), day -1, day 1 and 1 day before discharge
Prevalence of high PTH | Baseline (day -7), day -1, day 1 and 1 day before discharge
Prevalence of hypercalcemia | Baseline (day -7), day -1, day 1 and 1 day before discharge
Prevalence of hypomagnesemia | Baseline (day -7), day -1, day 1 and 1 day before discharge
30-day mortality | day 1 post-OP and 1 day before discharge
Clinical outcomes | day 1 post-OP and 1 day before discharge
  Including level of C-reactive protein and white blood cell (WBC) count
Complications after surgery | day 1 post-OP and 1 day before discharge
  Including in-hospital infectious complications, Dindo-Clavien classification, volume of ascites, duration of ascites, intra-abdominal abscess, postoperative haemorrhage, pleural effusion, wall abscess, and eventration.